CLINICAL TRIAL: NCT05217225
Title: The Association Between Parental Anxiety and Child Behavior During Simple Restorative Treatment: A Cross-Sectional Study.
Brief Title: The Association Between Parental Anxiety and Child Behavior.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farah Magdy Ramsis Farah Guirgis, Doctor, Cairo University
Other Study IDs: Child Behavior
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Parental Anxiety,Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Simple restorative treatment — Simple Occlusal Cavity class I then followed by final restoration

SUMMARY:
Parents' dental anxiety is demonstrated as a significant indicator for children's dental anxiety and parents play a key role in children's anxiety and fear development.

Studies have shown that parents who are fearful and anxious about dental treatments are associated with an increase in the occurrence of caries disease in their children, since they are more resistant to accompany their children to the dentist.

People with a high level of dental anxiety, both children and adults, can be difficult to treat, take longer, and have behavioral issues, all of which can lead to a stressful and unpleasant experience for both the patient and the dental practitioner

ELIGIBILITY:
Inclusion Criteria:

* Children, age ranging from 4 to 6 years old, of both sexes, have simple Occlusal cavities attending the pediatric dental clinic.
* Parents of both genders

Exclusion Criteria:

* Children who do not have the cognition to respond to the anxiety test or are not authorized by parents and medically compromised children.
* Parents who could not respond to the research tools.

Ages: 4 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: Children and parents attending to diagnosis clinics in Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Egypt.
Sampling Method: Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2022-06-24 (Estimated); Primary Completion 2022-10-24 (Estimated); Study Completion 2023-03-24 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Parental anxiety | baseline
  The Modified Dental Anxiety Scale Scores (5-25)

SECONDARY OUTCOMES:
Prevalence of Child Anxiety | Baseline
  The Modified Venham Picture Test Scores (0- 8)
Child behavior in dental care | During the procedure
  Venham Behavior Rating Scale.

IPD SHARING:
Plan to Share IPD: Undecided